CLINICAL TRIAL: NCT04445324
Title: Effects of Online and Recovery-oriented Peer Support Groups Facilitated by Peer Support Workers in Times of COVID-19 : A Feasibility Study of a Trial
Brief Title: Effects of Online and Recovery-oriented Peer Support Groups Facilitated by Peer Support Workers in Times of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Jean-Francois Pelletier, Associate Professor, Dpt of Psychiatry and Addictologye, University of Montreal, Centre de Recherche de l'Institut Universitaire en santé Mentale de Montréal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-2281
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Psychotic Disorders; Anxiety Depression
MeSH Terms: conditions — Psychotic Disorders | interventions — Control Groups

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional Online Peer Support Group (n=20) (Experimental): Trained Peer Support Workers (PSWs) from the Quebec Association of PSWs will organize and facilitate two series (one per condition) of 10 co-learning recovery workshops in a manner to simulate a typical peer support group. The difference of these transitional peer support groups to real community-based peer support groups is that (A) they will be facilitated by trained PSW, (B) they will have a personal-civic recovery focus, and (C) they will have a fixed, predetermined duration (10 weekly 60 to 90-minute online workshops). Typical Peer support groups bring together people who have similar concerns so they can explore solutions to overcome shared challenges and feel supported by others with similar experiences and who may better understand each other's situation. Peer support groups should ideally be independent from mental health and social services, although some services may facilitate and encourage the creation of (transitional) peer support groups, as is the case here. (WHO)
  Interventions: Behavioral: Transitional Online Peer Support Group (n=20); Other: Control Group (pharmacotherapy and/or psychotherapy, n=10)
- Control Group (pharmacotherapy and/or psychotherapy N=10) (Active Comparator): When individuals show up at the Emergency Department (T1) of the Montreal Mental Health University Institute, they are evaluated by the Evaluation and Liaison Module during their hospital stay when they are hospitalized. A diagnostic is established or confirmed by psychiatrists on the ward, and coded according to the World Health Organisation International Classification of Disease (ICD-10). According to these diagnoses, after discharge (T2) they are referred to a specialized outpatient clinic for an appointment (T3). Whether for (a) psychotic disorders or for (b) anxiety and mood disorders, pharmacotherapy or psychotherapy, or a combination of both, are then offered in accordance with guidelines of the Royal College of Physicians and Surgeons of Canada.
  Interventions: Other: Control Group (pharmacotherapy and/or psychotherapy, n=10)

INTERVENTIONS:
Behavioral: Transitional Online Peer Support Group (n=20) — Trained Peer Support Workers (PSWs) from the Quebec Association of PSWs will organize and facilitate two series (one per condition) of 10 co-learning recovery workshops in a manner to simulate a typical peer support group. The difference of these transitional peer support groups to real community-based peer support groups is that (A) they will be facilitated by trained PSW, (B) they will have a personal-civic recovery focus, and (C) they will have a fixed, predetermined duration (10 weekly 60 to 90-minute online workshops). Typical Peer support groups bring together people who have similar concerns so they can explore solutions to overcome shared challenges and feel supported by others with similar experiences and who may better understand each other's situation. Peer support groups should ideally be independent from mental health and social services, although some services may facilitate and encourage the creation of (transitional) peer support groups, as is the case here. (WHO)
  Arms: Transitional Online Peer Support Group (n=20)
Other: Control Group (pharmacotherapy and/or psychotherapy, n=10) — When individuals show up at the Emergency Department (T1) of the Montreal Mental Health University Institute, they are evaluated by the Evaluation and Liaison Module during their hospital stay when they are hospitalized. A diagnostic is established or confirmed by psychiatrists on the ward, and coded according to the World Health Organisation International Classification of Disease (ICD-10). According to these diagnoses, after discharge (T2) they are referred to a specialized outpatient clinic for an appointment (T3). Whether for (a) psychotic disorders or for (b) anxiety and mood disorders, pharmacotherapy or psychotherapy, or a combination of both, are then offered in accordance with guidelines of the Royal College of Physicians and Surgeons of Canada.

SUMMARY:
In times of pandemics, social distancing, isolation and quarantine exacerbate depression and anxiety as confined people are detached from their loved ones, deprived of personal liberties, and devoid of purpose owing to altered routine and livelihood (1,2). Those with pre-existing mental health problems or illnesses (MHPIs) might suffer from limiting interpersonal interactions that are central to their self-management, as well as reduced access to helpful but "non-essential" (often cancelled) psychiatric services (3). In response to this situation, this feasibility study of a trial consists of offering a transitional measure of online peer support for people suffering from (a) psychotic disorders or (b) anxiety and mood disorders, and to determine an effect size to this Peer Support Workers-delivered intervention in terms of both personal-civic recovery and clinical recovery (4). Peer Support Workers (PSWs) are persons with first-hand lived experience of MHPIs, and who are further along in their own recovery journey. As recommended by recovery-oriented best practices guidelines (5,6), upon training and certification they can provide supportive services when hired to fill such a paid specialty position directly in, or in conjunction with, current psychiatric services. Indeed, recovery focuses on how individuals can have more active control over their lives (agency). It is characterized by a search for the person's strengths and capacities, satisfying and meaningful social roles, and mobilizing formal and informal support systems. Peer support has thus become one predominant concept in the recovery paradigm and PSWs are specialized in peer support. Yet, not much is known about the efficacy of PSWs from a consumer's perspective of personal-civic recovery.

The five principal research questions are whether this online intervention will have an impact in terms of (Q1) personal-civic recovery potential and (Q2) clinical recovery potential, (Q3) how these potentials can be impacted by the COVID-19 pandemic, (Q4) how the lived experience of people in recovery can be mobilized to cope with such a situation, and (Q5) how sex and gender considerations can be taken into account for the pairing of PSWs with service users, beyond considerations based solely on psychiatric diagnoses or specific MHPIs.

DETAILED DESCRIPTION:
The "signatures" of MHPIs is a term formulated by the American National Institute of Mental Health to designate the broad range of genetic, biological, psychological, and social factors that may "sign" a specific mental disorder, depending on an individual's sex, history, lifestyle habits, and so on. In 2010, the Research Centre of the Montreal Mental Health University Institute (MMHUI), in Canada, implemented the "Signature Bank" project for the collection of biological and psychosocial dimensional signatures from all psychiatric emergency patients of the MMHUI (catchment area of about 600,000 inhabitants). More than 4,000 patients are treated annually at the MMHUI, while an additional 2,000 patients per year are treated by means of outpatient or ambulatory services. Our activities provide us with one of the largest populations of patients with MHPIs in Canada. By collaborating with the MMHUI Research Centre, MMHUI-hospital managers have contributed to the implementation of this large-scale project that aims at measuring the (epi)genetic, biological, psychological, and social signatures of people living with MHPIs who receive the MMHUI's clinical services. Typically, these measures are obtained at four different points in the clinical visit of patients at the MMHUI: (T1) when patients are admitted to the psychiatric emergency services, (T2) when they are discharged from the hospital, (T3) when they are admitted to an outpatient clinic, and (T4) 12 months after T3. This study now goes even further in understanding not only the signature of MHPIs, but also the dimensions of personal-civic recovery and as reported by our patients who will additionally complete the Recovery Assessment Scale (7), the Citizenship Measure (8) and the COVID19 Stress Scales (9) components.

Several instruments have been developed by clinicians and academics to assess clinical recovery. Based on their life narratives and to assess personal-civic recovery, measurement tools have also been developed through community-based participatory research and validated by persons living with MHPIs; for instance the Recovery Assessment Scale and the Citizenship Measure questionnaires. As users of mental health services typically tend to prefer interventions to help them recover, reintegrate with society, and achieve their personal goals, this pre-post research feasibility trial design is undertaken to evaluate the outcomes on personal-civic recovery (primary outcome) and on clinical recovery (secondary outcome). Among the Signature Bank participants diagnosed with (a) psychotic disorders, or (b) anxiety and mood disorders, and who have further accepted to be invited to participate in this study, an half will only receive the corresponding control intervention, and the other half will also receive our experimental Peer Support Workers' online group intervention based on peer support (random allocation control/experimental intervention ratio = 2:1). The abovementioned additional measures of personal-civic recovery and the COVID19 Stress Scales will be repeated, along with the measures of clinical recovery, which are routinely collected among all Signature Bank participants.

The aim is to collect data for a future Randomized Controlled Trial design by clarifying a certain number of remaining uncertainties and by determining an effect size that would be specifically attributable to transitional online peer support groups as facilitated by trained PSWs. Analyses will thus also consider scientific reasons, processes, resources, and management in preparation for a more definitive trial. Indicators of feasibility will include recruitment rates practices, participants and facilitators, as well as feasibility and retention rates in study protocol.

When a person shows up at the Emergency Department of MMHUI for the first time, he or she is systematically approached by a Research Nurse after a first medical authorization is granted for that person to be approached (sometimes this authorization is not granted for medical or security reasons). The Research Nurse then explains what objectives of the Signature Bank project are and invites the person to participate. Those who accept sign the Information and Consent Form (T1), fill out a series of questionnaires, including for sociodemographic information, consent to the taking of biological samples, and they are also asked if they accept to be contacted for other research purposes (like our own study). Then, as with any other MMHUI patients, they are evaluated by the Evaluation and Liaison Module during their hospital stay when they are hospitalized. A diagnostic is established or confirmed by psychiatrists on the ward, and coded according to the World Health Organisation International Classification of Disease (ICD-10). According to these diagnoses, after discharge (T2) they are referred to a specialized outpatient clinic (T3). Whether for psychotic disorders or for anxiety and mood disorders, pharmacotherapy or psychotherapy, or a combination of both, are then offered in accordance with guidelines of the Royal College of Physicians and Surgeons of Canada.

PSWs will learn with participants via a series of co-learning workshops that they will organize and facilitate as focus group panels in a manner to simulate a typical peer support group. The difference of our experimental and transitional online peer support groups to real community-based peer support groups is that (A) they will have to be facilitated by trained PSWs and (B) they will have a personal-civic recovery focus. They will also (C) have a fixed, predetermined duration (a series of 10 weekly 90-minute online workshops), and this is why they are said to be transitional. Indeed, as defined by the World Health Organization: "Peer support groups bring together people who have similar concerns so they can explore solutions to overcome shared challenges and feel supported by others who have had similar experiences and who may better understand each other's situation. Peer support groups may be considered by group members as alternatives to, or complementary to, traditional mental health services. They are run by members for members so the priorities are directly based on their needs and preferences. Peer support groups should ideally be independent from mental health and social services, although some services may facilitate and encourage the creation of peer support groups" (10).

The objective is to prevent the deterioration of the participants' recovery potential due to the COVID-19 pandemic and its aftermath. It is also about stimulating this potential by encouraging them to share their worries and their coping strategies in relation to the current situation. More generally, they will be asked to project themselves beyond this situation and to discuss future challenges of social inclusion and civic participation, for example by attending already existing community-based peer support groups, in the medium or long terms, and of which they will have heard of during the intervention. This is why this intervention is said to be transitional. Their own goals during the pandemic may be different from those post-pandemic and the effects of the response may also be different. However, the whole online intervention is intentionally designed to be readily adaptable to other (pandemic) situations.

To generate a collective narrative, the output of each workshop will be a brief written account of the group discussion, to which the next workshop will open up, and so on. To trigger discussion, PSWs will use animation cards and techniques inspired and adapted from materials initially designed to help healthcare teams develop the psychosocial skills of patients in Therapeutic Patient Education. Each workshop will be filmed via a secured video communication system for subsequent qualitative observational and content analyses. In accordance with our model of patient engagement, PSWs will each time start by disclosing being themselves persons in recovery, and feed with content drawn from their lived experience while asking participants to share their own lived experience and coping strategies. This is in line with experiential learning (11). After each workshop, the PSWs will meet for a 30-minute debriefing session, asking themselves what they have just learned, personally and professionally (also recorded). This is a process of recovery mentorship as an expression of psychological empowerment, as embodied in and practiced by the PSWs as mentors, and as an egalitarian relation that helps facilitate the empowerment of the mentees (12).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with (1) schizophrenia and psychotic disorders (ICD F20-F29), or
* Patients diagnosed with (2) anxiety or mood disorders (ICD F30-F49)

Exclusion Criteria:

* Active suicidal intentions
* Marked cognitive impairment
* No access to an electronic device with a webcam and microphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of patients' current status : recovery (personal recovery) | 14 weeks
  Recovery Assesment Scale (RAS). This is a 24-item questionnaire with 5-point Likert scales (1-2-3-4-5). Higher scores are positively correlated with higher levels of recovery. Minimum score = 24 : maximum score = 120.
Assessment of patients' current status : citizenship (personal recovery) | 14 weeks
  Participating patients will fill out the Citizenship Measure (CM). This is a 23-item questionnaire with 5-point Likert scales (1-2-3-4-5). Higher scores are positively correlated with higher levels of citizenship. Minimum score = 23 : maximum score = 115.
Assessment of patients' current status : COVID-19 Stress Scales | 14 weeks
  Participating with 5-point Likert scales (0-1-2-3-4). Higher scores are positively correlated with higher levels of COVID-related levels of stress. Minimum score = 0 : maximum score = 144.

SECONDARY OUTCOMES:
Assessment of patients' current status : anxiety (clinical recovery) | 14 weeks
  Participating patients will fill out the Anxiety State-Trait Anxiety Inventory Form Y6 (STAI-Y6). This is a 6-item questionnaire with 4-point Likert scales (1-2-3-4). Higher scores are positively correlated with higher levels of anxiety. Minimum score = 6 : maximum score = 24.
Assessment of patients' current status : depression (clinical recovery) | 14 weeks
  Participating patients will fill out the Depression Patient Health Questionnaire (PHQ-9). This is a 9-item questionnaire with 4-point Likert scales (0-1-2-3). Higher scores are positively correlated with higher levels of depression. Minimum score = 0 : maximum score = 27.
Assessment of patients' current status : alcohol dependence (clinical recovery) | 14 weeks
  Participating patients will fill out the Alcohol Use Disorders Identification Test (AUDIT-10). This is a 10-item questionnaire with 5-point Likert scales (0-1-2-3-4). Higher scores are positively correlated with higher levels of alcohol dependence. Minimum score = 0 : maximum score = 40.
Assessment of patients' current status : drug dependence (clinical recovery) | 14 weeks
  Participating patients will fill out the Drug Abuse Screening Test (DAST-10). This is a 10-item questionnaire with noyes answers (0-1). Higher scores are positively correlated with higher levels of drog dependence. Minimum score = 0 : maximum score = 10.
Assessment of patients' current status : psychosis (clinical recovery) | 14 weeks
  Psychosis Screening Questionnaire (PSQ 12 items) with no-unsure-yes answers (1-2-3). Higher scores are positively correlated with higher levels of psychosis. Minimum score = 12 : maximum score = 36.
Assessment of patients' current status : social functioning (clinical recovery) | 14 weeks
  Participating patients will fill out the World Health Organization Disability Assessment Schedule (WHODAS 2.0). This is a 12-item questionnaire with 5-point Likert scales (0-1-2-3-4). Lower scores are positively correlated with higher levels of social functioning. Minimum score = 0 : maximum score = 48.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Pelletier, PhD, Principal Investigator — Research Centre - Montreal Mental Health University Institute
Locations (1):
- CR-IUSMM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelletier JF, Houle J, Goulet MH, Juster RP, Giguere CE, Bordet J, Henault I, Lesage A, De Benedictis L, Denis F, Ng R. Online and Recovery-Oriented Support Groups Facilitated by Peer Support Workers in Times of COVID-19: Protocol for a Feasibility Pre-Post Study. JMIR Res Protoc. 2020 Dec 18;9(12):e22500. doi: 10.2196/22500. PMID 33259326
- See also: 1 . Hawryluck, L., Gold, W. L., Robinson, S., Pogorski, S., Galea, S., & Styra, R. (2004). SARS control and psychological effects of quarantine, Toronto, Canada. Emerging infectious diseases, 10(7), 1206-1212. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3323345/
- See also: 2. Jeong, H., Yim, H. W., Song, Y. J., Ki, M., Min, J. A., Cho, J., & Chae, J. H. (2016). Mental health status of people isolated due to Middle East Respiratory Syndrome. Epidemiology and health, 38, e2016048. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5177805/
- See also: 3. Venkatesh Ashwin, Edirappuli Shantal. (2020) Social distancing in covid-19: what are the mental health implications? BMJ 2020; 369 :m1379 — https://pubmed.ncbi.nlm.nih.gov/32253182/
- See also: 4. Pelletier JF, Corbière M, Lecomte T, Briand C, Corrigan P, Davidson L, Rowe M. (2015) Citizenship and recovery: two intertwined concepts for civic-recovery. BMC Psychiatry. 2015;15(37):1-7. — https://pubmed.ncbi.nlm.nih.gov/25885779/
- See also: 5. van Vugt M, Kroon H, Delespaul P, Mulder C. (2012). Consumer-Providers in Assertive Community Treatment Programs: Associations With Client Outcomes. Psychiatr Serv. 2012;63(5):477-81. — https://pubmed.ncbi.nlm.nih.gov/22388475/
- See also: 6. Mental Health Commission of Canada. (2015). Guidelines for Recovery-Oriented Practice — https://www.mentalhealthcommission.ca/sites/default/files/MHCC_RecoveryGuidelines_ENG_0.pdf
- See also: 7. Corrigan PW, Salzer M, Ralph RO, Sangster Y, Keck L. Examining the Factor Structure of the Recovery Assessment Scale. Schizophr Bull. 2004;30(4):1035-41. — https://pubmed.ncbi.nlm.nih.gov/15957202/
- See also: 8. Rowe M, Clayton A, Benedict P, Bellamy C, Antunes K, Miller R, Pelletier, JF al. Going to the Source: Creating a Citizenship Outcome Measure by Community-Based Participatory Research Methods. Psychiatr Serv. 2012;63(5):445-50. — https://pubmed.ncbi.nlm.nih.gov/22549531/
- See also: 9. Taylor, S., Landry, C. A., Paluszek, M. M., Fergus, T. A., McKay, D., & Asmundson, G. (2020). Development and initial validation of the COVID Stress Scales. Journal of anxiety disorders, 72, 102232. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7198206/
- See also: 10. Peer support groups by and for people with lived experience. WHO QualityRights guidance module. Geneva: World Health Organization; 2019. — https://apps.who.int/iris/handle/10665/329644
- See also: 11. Yardley S, Teunissen P, Dornan T. Experiential learning: transforming theory into practice. Med Teach. 2012;34(2):161-164. — https://pubmed.ncbi.nlm.nih.gov/22288996/
- See also: 12. Christens, B. D. Toward relational empowerment. American Journal of Community Psychology. 2012;50(1-2):114-28. — https://pubmed.ncbi.nlm.nih.gov/22094588/
- See also: STAI-Y-short: Marteau TM, Bekker H. The development of a six-item short form of the state scale of the Spielberger State - Trait Anxiety Inventory (STAI). British Journal of Clinical Psychology. 1992;31:301-306. — https://pubmed.ncbi.nlm.nih.gov/1393159/
- See also: PHQ-9: Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. Journal of General Internal Medicine. 2001;16:606-13. — https://pubmed.ncbi.nlm.nih.gov/11556941/
- See also: AUDIT: Babor et al. The AUDIT guidelines for use in primary care. 2nd ed. World Health Organization. 2001. — https://apps.who.int/iris/handle/10665/67205
- See also: DAST-10: Lam, L. P., Leung, W. C., Ip, P., Chow, C. B., Chan, M. F., Ng, J. W. Y., … Chin, R. K. H. Validation of the Drug Abuse Screening Test (DAST-10): A study on illicit drug use among Chinese pregnant women. Scientific Reports. 2015;5, 11420. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4473689/
- See also: PSQ: Bebbington PE, Nayani T. The Psychosis Screening Questionnaire. International Journal of Methods in Psychiatric Research. 1995;5: 11-19. — https://www.scirp.org/journal/paperinformation.aspx?paperid=62317
- See also: WHODAS : Federici S, Bracalenti M, Meloni F, Luciano JV. World Health Organization disability assessment schedule 2.0: An international systematic review. Disabil Rehabil. 2017;39(23):2347-2380. — https://pubmed.ncbi.nlm.nih.gov/27820966/